CLINICAL TRIAL: NCT00030173
Title: A Phase 1, Dose Escalation Trial to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Epothilone D in Patients With Advanced Solid Tumors
Brief Title: A Trial to Evaluate Epothilone D in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KOS-101; NCT00033501 (obsolete NCT alias)
Record Dates: First submitted 2002-02-07; First posted 2002-02-08 (Estimated); Last update posted 2009-01-08 (Estimated); Status verified 2009-01

CONDITIONS: Neoplasms
Keywords: Epothilone D; tubulin polymerization
MeSH Terms: conditions — Neoplasms | interventions — desoxyepothilone B

INTERVENTIONS:
Drug: Epothilone D (KOS-862)

SUMMARY:
Epothilone D represents one of a class of cytotoxic macrolides capable of causing mitotic arrest by stabilizing tubulin polymerization. Since microtubules are essential for mitosis, motility, secretion and proliferation, the observed antitumor effects of epothilones have been attributed to their ability to initiate cell death by inhibiting such processes. Epothilone D has demonstrated in vitro cytotoxic activity in a panel of human cell lines, equipotent to that of paclitaxel. In vivo, Epothilone D has also shown significant antitumor activity in a range of xenograft models, including paclitaxel-resistant xenografts. Epothilone D is more potent than paclitaxel in cell lines that demonstrate multiple drug resistant activity overexpressing p-glycoprotein.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of histologically documented, advanced stage, primary or metastatic adult solid tumors that are refractory to standard therapy or for which no curative standard therapy exists. This includes but is not limited to cancers of the breast, ovary, head and neck, esophagus, lung, gastrointestinal tract, and sarcomas.
2. Evidence of radiographically measurable or evaluable disease.

Exclusion Criteria:

1. Pre-existing peripheral neuropathy of CTC Grade > 2 due to any cause.
2. Documented hypersensitivity reaction (CTC Grade > 2) to prior paclitaxel or other therapy containing Cremophor.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2001-10; Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- UCLA Medical Center, Los Angeles, California, United States